CLINICAL TRIAL: NCT06346327
Title: Clinical Significance Of Intermittently Absent End-Diastolic Flow Of The Fetal Umbilical Artery On Perinatal And Neonatal Outcomes Zeynep Kayaoğlu Yıldırım, Gynecologist and Obstetrician, Perinatologist, İstanbul Başakşehir Çam ve Sakura City Hospital, Drkayaoglu@Hotmail.Com, Alperen İnce, MD, Obstetrics and Gynecology Medical Student, Başakşehir Çam ve Sakura City Hospital,Gökhan Bayanmelek, Gynecologist and Obstetrician, Perinatologist, İstanbul Başakşehir Çam ve Sakura City Hospital,Gökhan Bolluk, Gynecologist and Obstetrician, Perinatologist, Başakşehir Çam ve Sakura City Hospital
Brief Title: Clinical Significance Of Intermittently Absent End-Diastolic Flow Of The Fetal Umbilical Artery On Perinatal And Neonatal Outcomes Dr. Zeynep Kayaoğlu Yıldırım Dr. Alperen İnce Dr Gökhan Bayanmelek Dr Gökhan Bolluk
Status: Completed | Type: Observational
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Zeynep Kayaoğlu Yıldırım, Gynecologist and Obstetrician, Perinatology fellow, Başakşehir Çam & Sakura City Hospital
Other Study IDs: Absent End-Diastolic Flow
Record Dates: First submitted 2024-03-16; First posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Absent End-Diastolic Flow Of The Fetal Umbilical Artery
Keywords: absent end-diastolic flow, Doppler, pregnancy outcome, neonatal outcomes, umbilical artery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Objective: This study aimed to estimate the risk of adverse perinatal outcomes among pregnant patients with intermittently absent (iAEDF) and persistently absent end-diastolic umbilical artery flow (pAEDF). The fetal risks associated with persistently absent end-diastolic flow have been described. However, the risks associated with intermittent absent end-diastolic flow are not well-known.

Study design: We performed a retrospective cohort study of patients diagnosed with the iAEDF or pAEDF at our institution from 2020 to 2023. Fetuses were classified under two categories: iAEDF group and pAEDF group.Neonatal outcomes, demographic information, pregnancy outcomes and pregnancy complications were compared between patients with iAEDF and those with pAEDF.

DETAILED DESCRIPTION:
Doppler velocity measurement of the umbilical artery (UA) serves as a crucial clinical tool for monitoring feto-placental hemodynamics and assessing fetal well-being in high-risk pregnancies. This technique has demonstrated notable advantages in monitoring potentially risky fetuses, particularly in pregnancies complicated by placental disorders, such as fetal growth restriction (FGR). Since UA Doppler (UAD) results can deteriorate over the course of pregnancy, regular assessments are recommended. However, the frequency of these assessments, management protocols, and delivery timing recommendations vary among major national obstetric societies.

The UA blood velocity waveform is typically characterized by the pulsatility index (PI) and qualitative information concerning the potential absence or reversal of end-diastolic flow (EDF). Absent end-diastolic flow (AEDF) signifies increased resistance to flow in the placental vascular bed and is associated with elevated risks of intrauterine death and adverse perinatal outcomes. AEDF in the UA can be either persistent (pAEDF), occurring in most or all fetal cardiac cycles, or intermittent (iAEDF), manifesting in only some of the cardiac cycles. However, standardized definitions for these terms lack and the clinical implications of the iAEDF versus the pAEDF remain unclear.

A previous study indicated that, compared to fetuses with pAEDF, those with iAEDF are diagnosed with UAD abnormalities later in pregnancy and are delivered at a later gestational age (GA) with higher birth weights. Consequently, it is plausible that some fetuses with an iAEDF may remain in utero for an extended duration without facing an immediate risk of death. Identifying this specific subgroup might allow the avoidance of some neonatal risks associated with extremely preterm birth.

In this study, we aimed to assess the risk of adverse perinatal outcomes among pregnant patients with intermittently absent and persistently absent end-diastolic umbilical artery flow. This investigation seeks to contribute to a better understanding of the fetal risks associated with different patterns of absent end-diastolic flow, thereby informing clinical management and decision-making for high-risk pregnancies.

We performed a retrospective cohort study of patients with non-anomalous, singleton pregnancies diagnosed with intermittent absence of end-diastolic umbilical artery Doppler flow or persistent absence of end-diastolic flow at our institution from 2020 to 2023. The study was approved by the Başakşehir Çam ve Sakura City Hospital Clinical Research Ethics Committee (ethics no.2023-561, date 08/11/2023) and was conducted in accordance with the latest version of the Declaration of Helsinki (2019/92). Fetuses were classified into two categories: intermittent absent end-diastolic flow and persistent absent end-diastolic flow.

Patients were excluded if they had major fetal anomalies or aneuploidy diagnosed prenatally or if they lacked delivery or neonatal outcome data. Patients were also excluded if they were intermittently elevated or if they showed REDF syndrome during pregnancy. All ultrasounds were performed and interpreted by a maternal-fetal medicine fellowship-trained obstetrician. UAD waveforms were obtained through transabdominal imaging from a free-floating loop of the umbilical cord on a Hitachi machine. To improve the accuracy of the measurements, waveforms were obtained during a brief pause during maternal breathing. At least three separate UAD assessments were performed for each fetus. Doppler waveforms were defined as iAEDF if diastolic flow was absent in one or more waveforms during a cycle of images. Doppler waveforms were defined as persistently absent if the absence of diastolic flow was observed in all waveforms. The REDF was defined as the reversal of flow in the UA in at least one fetal cardiac cycle. The patients defined as having an iAEDF were not subdivided based on the percentage of patients with no waveforms. The most recent guidelines for the management of FGR from the Society for Maternal-Fetal Medicine and American College of Obstetricians and Gynecologists (ACOG) were released in 2020. We recommend that pregnant patients with AEDF undergo UAD surveillance two to three times weekly and delivery by 33 to 34 weeks of gestation. Inpatient management is suggested as an option for AEDF. In our study, the management of AEDF included admission of pregnant patients for antenatal corticosteroid administration and inpatient monitoring, including daily UAD assessment and antenatal testing twice a day. Although previous studies have shown that improvements in UAD abnormalities can be observed with the application of corticosteroids to stimulate fetal lung maturity, we did not find it necessary to study it since corticosteroids were already administered to all patients whose AEDF was detected. Delivery was recommended at the GA of 34 weeks following the recommendations of ACOG, or if another indication arose. If a diagnosis of AEDF or REDF was made after the recommended GA for delivery, it was advised to proceed with delivery at the time of diagnosis.

Maternal demographic information, medical complications, prenatal history (including additional ultrasound studies), and delivery and neonatal outcomes were taken from medical records.

The primary outcome was a composite of neonatal outcomes including birth weight, Z-score for standardized birth weight, Apgar score in the first minute, Apgar score in the fifth minute, Apgar score in the fifth minute lower than seven, admission to the ICU and the need for intubation.

Demographic information, time of AEDF diagnosis, latency from the time of AEDF diagnosis to delivery, and pregnancy complications (IUMF, ablatio placenta, fetal distress, IUGR, amniotic fluid abnormalities) were the other outcomes.

These outcomes were compared between patients with iAEDF and those with pAEDF. Statistical Analysis Statistical analysis was performed using R statistical software (R Core Team 2021). A score of P<0.05 was considered to indicate statistical signiﬁcance. The normality of the distribution of the variables was assessed using quantile-quantile plots and the Shapiro-Wilk test. Continuous variables were evaluated using the unpaired student's t test or Mann-Whitney U test (for two groups), depending on the normality of the distribution. Categorical variables were analyzed using the χ2 test or Fisher's exact test, depending on the variable count.

ELIGIBILITY:
Inclusion Criteria:

- Pregnancies with absent umbilical artery end-diastolic velocity

Exclusion Criteria:

* Multiple pregnancies
* Pregnancies with unknown outcomes

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Singleton pregnancies with absent umbilical artery end-diastolic velocity between the ages of 18-45
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
neonatal outcomes | first 24 hours after birth
  The primary outcome was a composite of neonatal outcomes, including birth weight (weight in grams), Z-score for standardized birth weight (weight in grams), Apgar score in the first minute, Apgar score in the fifth minute, Apgar score in the fifth minute lower than seven, admission to the ICU, and the need for intubation.These outcomes were compared between patients with intermittantly absent end-diastolic flow and those with persistantly absent end-diastolic flow.
latency from the time of absent endiastolic flow diagnosis to delivery | time from diagnosis to birth
  time (time in days) elapsed from diagnosis to birth was compared between patients with iAEDF and those with pAEDF.
pregnancy complications (Number of Pregnancies complicated with IUMF, ablatio placenta, fetal distress, Intrauterine growth restriction and amniotic fluid abnormalities). | time from diagnosis to birth
  Pregnancy complications were compared between patients with iAEDF and those with pAEDF.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Kayaoğlu Yıldırım, MD, Principal Investigator — Çam ve Sakura City Hospital
Locations (1):
- İstanbul Başakşehir Çam ve Sakura City Hospital, Istanbul, Türkiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Green S, Schmidt A, Gonzalez A, Bhamidipalli SS, Rouse C, Shanks A. Clinical significance of intermittent absent end-diastolic flow of the umbilical artery in fetal growth restriction. Am J Obstet Gynecol MFM. 2023 Feb;5(2):100800. doi: 10.1016/j.ajogmf.2022.100800. Epub 2022 Nov 9. PMID 36371037
- [Background] Rosner J, Rochelson B, Rosen L, Roman A, Vohra N, Tam Tam H. Intermittent absent end diastolic velocity of the umbilical artery: antenatal and neonatal characteristics and indications for delivery. J Matern Fetal Neonatal Med. 2014 Jan;27(1):94-7. doi: 10.3109/14767058.2013.806475. Epub 2013 Jun 26. PMID 23682642
- [Background] Bligard KH, Xu X, Raghuraman N, Dicke JM, Odibo AO, Frolova AI. Clinical significance of umbilical artery intermittent vs persistent absent end-diastolic velocity in growth-restricted fetuses. Am J Obstet Gynecol. 2022 Sep;227(3):519.e1-519.e9. doi: 10.1016/j.ajog.2022.06.005. Epub 2022 Jun 10. PMID 35697096

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-08): https://cdn.clinicaltrials.gov/large-docs/27/NCT06346327/Prot_SAP_000.pdf